CLINICAL TRIAL: NCT05612828
Title: The Efficacy of Simulation Manikins in the Military Medics Training
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: VentRes-2022-01-JP
Record Dates: First submitted 2022-10-29; First posted 2022-11-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: War-Related Injuries
Keywords: Combat Life Saver; Simulation Medicine; Stress response
MeSH Terms: conditions — War-Related Injuries; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional training (Experimental): Combat Life Savers trained by conventional combat medicine approach.
  Interventions: Behavioral: Conventional versus simulation manikin training
- Simulation manikin training (Experimental): Training based on principles of simulation medicine.
  Interventions: Behavioral: Conventional versus simulation manikin training

INTERVENTIONS:
Behavioral: Conventional versus simulation manikin training — Two approaches to training Combat Life Savers will be employed and performance of participants will be evaluated.

SUMMARY:
The aim of the study is to verify the applicability of simulation manikin in combat training of military medics. The research will be conducted on healthy volunteers - medics of the Czech Armed Forces, as a part of the compulsory medical courses required for foreign military missions as a "Combat Life Saver". Comparison of the performance of two groups of course participants who were trained using the standard approach versus experiential learning using simulation manikins.

DETAILED DESCRIPTION:
With the development of modern hi-tech manikins and their growing popularity in the training of "civilian" medics, the possibilities of their application in the training of military medics are emerging. The aim of the study is to verify the applicability of simulation manikin in combat training of military medics. The research will be conducted on healthy volunteers - medics of the Czech Armed Forces, as a part of the compulsory medical courses required for foreign military missions as a "Combat Life Saver". Comparison of the performance of two groups of course participants who were trained using the standard approach versus experiential learning using simulation manikins. In addition to monitoring the particular professional performance of the trainees, changes in basic physiological functions, including the endocrinological response to stress conditions, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* active soldier during the Tactical Combat Casualty Care course

Exclusion Criteria:

* not willing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration time of the of use of tourniquet | 10 minutes
  Time to complete diagnostics and treatment of bleeding (in seconds)
Correctness of treatment of severe bleeding | 10 minutes
  Based on standardized forms (points on a standardised scale)
Duration time of the of use of nasal airway | 10 minutes
  Time to complete diagnostics and treatment of airway obstruction (in seconds)
Correctness of treatment of airway obstruction | 10 minutes
  Based on standardized forms (points on a standardised scale)
Duration time of the use of chest seal | 10 minutes
  Time to complete diagnostics and treatment of open pneumothorax (in seconds)
Correctness of treatment of open pneumothorax | 10 minutes
  Based on standardized forms (points on a standardised scale)

SECONDARY OUTCOMES:
Stress level 1 | 1 hour
  Level of stress response based on changes in blood pressure (in mm of mercury)
Stress level 2 | 1 hour
  Level of stress response based on changes in heart rate (in beats per minute)
Stress level 3 | 1 hour
  Level of stress response based on changes in cortisol level (in nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubík, Ph.D., Study Director — Czech Technical University in Prague
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: upon final publication
Access Criteria: open access
URL: https://ventilation.fbmi.cvut.cz/data/

REFERENCES:
- [Background] McCarthy M. US military revamps combat medic training and care. Lancet. 2003 Feb 8;361(9356):494-5. doi: 10.1016/S0140-6736(03)12494-4. No abstract available. PMID 12583953